CLINICAL TRIAL: NCT00219661
Title: Impact of Drainage of Subglottic Secretions on Ventilator-Associated Pneumonia:a Randomised Multicentre Trial
Brief Title: Effect of Drainage of Subglottic Secretions on Pneumonia Acquired Under Mechanical Ventilation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Poissy-Saint Germain Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 323
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2007-04-23 (Estimated); Status verified 2007-04

CONDITIONS: ICU's Patients Under Mechanical Ventilation
Keywords: randomised control trial; intensive care unit; mechanical ventilation; ventilator-associated pneumonia; drainage of subglottic secretions
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: drainage of subglottic secretions (HiLo Evac tube)

SUMMARY:
The purpose of this study is to determine whether drainage of subglottic secretions is effective to reduce the incidence of pneumonia acquired under mechanical ventilation in ICU's patients.

DETAILED DESCRIPTION:
Nosocomial infection represent a major problem in hospitals. In intensive care units, ventilator-associated pneumonia (VAP) is associated with an increase in morbidity and mortality. Incidence of VAP is high, 20 to 30% of patients under mechanical ventilation (MV) for more than 48 hours. In the pathogenesis of VAP, two processes are considered essential for its development: bacterial colonization of the oropharynx and tracheobronchial tract, followed by aspiration of contaminated secretions into the lower airways. It has been shown that pooled secretions above inflated endotracheal tube cuffs may be source of aspiration and can be a cause of VAP. Several studies have suggested that recurrent aspiration of subglottic secretions can be prevented by intermittent drainage of subglottic secretions. Nevertheless, recent CDC guideline reported that there was not enough evidence to conclude on the efficacy of such intervention.

During the study, patients, in both groups, will be intubated with the same device permitting subglottic drainage (HiLo Evac endotracheal tube). The daily screening of VAP will be performed until the 28th days of mechanical ventilation without occurrence of VAP. The follow-up of each patient will be realized until the ICU's discharge.

Comparison: The incidence of VAP will be compared between two groups: one group with intermittent drainage of subglottic secretions and the other one without this intervention.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients expected to require MV more than 48 hours

Exclusion Criteria:

* patients already intubated for more than 12 hours
* patients intubated with another tube than the HiLo Evac tube
* patients admitted for cardiac arrest
* patients admitted for self poisoning
* patients admitted with tracheotomy
* patients already included in an another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440
Dates: Start 2003-06; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Incidence of ventilator-associated pneumonia(VAP)

SECONDARY OUTCOMES:
Duration on mechanical ventilation (MV)
Prior duration of MV before occurrence of VAP
duration of ICU's stay
Rate of tracheotomy
ICU's mortality
Microbiology of the VAP

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Lacherade, M.D., Principal Investigator — Medical Intensive Care Unit, Poissy-Saint-Germain Hospital
Locations (4):
- France (4):
  - Avignon Hospital, Avignon
  - André Mignot Hospital, Le Chesnay
  - Poissy Saint-Germain Hospital, Poissy
  - Poisyy Saint-Germain Hospital, Saint-Germain-en-Laye

REFERENCES:
- [Derived] Lacherade JC, De Jonghe B, Guezennec P, Debbat K, Hayon J, Monsel A, Fangio P, Appere de Vecchi C, Ramaut C, Outin H, Bastuji-Garin S. Intermittent subglottic secretion drainage and ventilator-associated pneumonia: a multicenter trial. Am J Respir Crit Care Med. 2010 Oct 1;182(7):910-7. doi: 10.1164/rccm.200906-0838OC. Epub 2010 Jun 3. PMID 20522796